CLINICAL TRIAL: NCT00821678
Title: Telemedicine Outreach for Post Traumatic Stress in CBOCs
Acronym: TOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI 08-098
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: telemedicine; rural; veterans; care management; psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Telemedicine Outreach for PTSD (Experimental): Telemedicine-Based Collaborative Care
  Interventions: Other: Telemedicine Outreach for PTSD
- Arm 2 Treatment as usual (No Intervention): Usual Care

INTERVENTIONS:
Other: Telemedicine Outreach for PTSD — The intervention involves an off-site PTSD care team (tele-psychiatrist, tele-psychologist, tele-pharmacist, and tele-nurse care manager) and uses telemedicine technologies (telephone, interactive video and electronically shared medical records). A dedicated nurse telephone care manager educates/activates patients, identifies preferences, overcomes treatment barriers, monitors symptoms, side-effects and adherence, identifies psychiatric comorbidities, and encourages patient self-management. Tele-pharmacists provide medication management by phone. Tele-psychologists provide Cognitive Processing Therapy via interactive video. Tele-psychiatrists supervise the off-site care team as well as conduct consultations and provide medication management via interactive video.
  Other Names: Telemedicine-Based Collaborative Care
  Arms: Arm 1 Telemedicine Outreach for PTSD

SUMMARY:
The purpose of this study is improved outcomes for veterans with Post Traumatic Stress Disorder (PTSD) treated in small VA Community Based Outpatient Clinics (CBOCs). Although psychotherapy and pharmacotherapy treatments for PTSD have been proven to be efficacious in controlled trials, geographic barriers often prevent veterans from accessing these evidence-based treatments. Telemedicine technologies will be used to overcome geographic barriers to care. Specifically, we will evaluate the Telemedicine Outreach for PTSD (TOP) intervention which is based on the principals of the Chronic Care Model and Disease Management, and builds on the evidence base of quality improvement for depression in primary care settings. The TOP intervention will employ an off-site PTSD care team (tele-psychiatrist, tele-psychologist, tele-pharmacist, and tele-nurse care manager) and will use telemedicine technologies (telephone, interactive video and electronically shared medical records) to treat CBOC patients with a newly emerging or chronic PTSD. We hypothesize that study participants randomized to the TOP intervention will receive higher quality of care and experience better outcomes compared to study participants randomized to treatment as usual.

DETAILED DESCRIPTION:
Approximately 400 Veterans with PTSD will be recruited from nine CBOCs in VISN 16 and 22. Veterans screening positive for PTSD and those already in active treatment will be recruited. Patients actively engaged in specialty PTSD treatment at the parent VAMC will be excluded. Patients will be the unit of randomization. A dedicated nurse telephone care manager will educate/activate patients, identify treatment preferences, overcome treatment barriers, monitor symptoms, side-effects and adherence, identify psychiatric comorbidities, and encourage patient self-management. Tele-pharmacists will provide medication management by phone. Tele-psychologists will provide Cognitive Processing Therapy (without exposure) via interactive video. Tele-psychiatrists will supervise the off-site care team as well as conduct consultations and provide medication management via interactive video. Telephone interviews will be administered at baseline, six and twelve months by blinded research assistants. Process of care measures will include: 1) whether the veteran received a documented treatment concordant with VA/DoD PTSD Treatment Guidelines, 2) self-reported adherence to treatment, and 3) satisfaction with care as measured by Experience of Care and Health Outcomes (ECHO) Survey. Clinical outcomes will include: 1) PTSD severity as measured by the Posttraumatic Diagnostic Scale (PDS), 2) depression severity as measured by the PHQ9, 3) quantity and frequency of alcohol consumption, 4) health status as measured by the SF12V and 5) quality of life as measured by the Quality of Well-Being (QWB) scale. Activity based costing methods will be used to measure intervention cost data.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic Criteria for PTSD (CAPS),
* veterans,
* treated in CBOC

Exclusion Criteria:

* schizophrenia,
* bipolar disorder,
* current substance dependence,
* current specialty PTSD treatment at VA Medical Center,
* no access to telephone,
* hearing or speech impediment,
* terminal illness,
* non-capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fortney, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System (North Little Rock), North Little Rock, Arkansas
  - VA Medical Center, Loma Linda, Loma Linda, California
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana

REFERENCES:
- [Result] Fortney JC, Pyne JM, Kimbrell TA, Hudson TJ, Robinson DE, Schneider R, Moore WM, Custer PJ, Grubbs KM, Schnurr PP. Telemedicine-based collaborative care for posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Jan;72(1):58-67. doi: 10.1001/jamapsychiatry.2014.1575. PMID 25409287
- [Result] Grubbs KM, Fortney JC, Pyne JM, Hudson T, Moore WM, Custer P, Schneider R, Schnurr PP. Predictors of Initiation and Engagement of Cognitive Processing Therapy Among Veterans With PTSD Enrolled in Collaborative Care. J Trauma Stress. 2015 Dec;28(6):580-4. doi: 10.1002/jts.22049. PMID 26625355
- [Result] Grubbs KM, Fortney JC, Kimbrell T, Pyne JM, Hudson T, Robinson D, Moore WM, Custer P, Schneider R, Schnurr PP. Usual Care for Rural Veterans With Posttraumatic Stress Disorder. J Rural Health. 2017 Jun;33(3):290-296. doi: 10.1111/jrh.12230. Epub 2017 Jan 23. PMID 28112433
- [Result] Painter JT, Fortney JC, Austen MA, Pyne JM. Cost-Effectiveness of Telemedicine-Based Collaborative Care for Posttraumatic Stress Disorder. Psychiatr Serv. 2017 Nov 1;68(11):1157-1163. doi: 10.1176/appi.ps.201600485. Epub 2017 Jul 3. PMID 28669290
- [Derived] Campbell SB, Erbes C, Grubbs K, Fortney J. Social Support Moderates the Association Between Posttraumatic Stress Disorder Treatment Duration and Treatment Outcomes in Telemedicine-Based Treatment Among Rural Veterans. J Trauma Stress. 2020 Aug;33(4):391-400. doi: 10.1002/jts.22542. Epub 2020 Jun 10. PMID 32521100

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Telemedicine Outreach for PTSD: Telemedicine-Based Collaborative Care
  Telemedicine Outreach for PTSD: The Telemedicine Outreach for PTSD (TOP) intervention will employ an off-site PTSD care team (tele-psychiatrist, tele-psychologist, tele-pharmacist, and tele-nurse care manager) and will use telemedicine technologies (telephone, interactive video and electronically shared medical records). A dedicated nurse telephone care manager will educate/activate patients, identify treatment preferences, overcome treatment barriers, monitor symptoms, side-effects and adherence, identify psychiatric comorbidities, and encourage patient self-management. Tele-pharmacists will provide medication management by phone. Tele-psychologists will provide Cognitive Processing Therapy (without exposure) via interactive video. Tele-psychiatrists will supervise the off-site care team as well as conduct consultations and provide medication management via interactive video.
- Arm 2 Treatment as Usual: Treatment as usual
Period: Overall Study
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Started | 133 | 132
Completed | 112 | 118
Not Completed | 21 | 14
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Lost to Follow-up | 13 | 12
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual | Total
Number analyzed (Participants) | 133 | 132 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (14.0) | 52.5 (13.6) | 52.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 118 | 120 | 238
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian Non-Hispanic | 77 | 92 | 169
  Caucasian Hispanic | 12 | 8 | 20
  African American | 31 | 21 | 52
  Other Race/Ethnicity | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptom Severity (PDS)
Description: range - 0-51 (higher score represents greater severity)
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 112 | 118
units on a scale | -5.31 (10.91) | -1.07 (7.73)
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Slope = -3.81, 95% CI 2-sided [-6.19 to -1.43]

2. Secondary Outcome: Change in Continuous Measure of Depression Symptom Severity (SCL-20)
Description: range - 0-4 (higher score represents greater severity
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 112 | 118
units on a scale | -0.43 (0.62) | -0.16 (0.56)
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Slope = -0.25, 95% CI 2-sided [-0.4 to -0.1]

3. Secondary Outcome: Change in Continuous Measure of Alcohol Use (Audit Score)
Description: range - 0-12 (higher score represents greater severity)
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 112 | 118
units on a scale | -0.36 (2.19) | -0.17 (1.73)
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.33 to 0.70]

4. Secondary Outcome: Change in Continuous Measure of Health Status (SF12V PCS)
Description: range - 0-100 (higher score represents greater physical health status)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 112 | 118
units on a scale | 0.77 (7.50) | -1.45 (9.47)
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Slope = 2.67, 95% CI 2-sided [0.45 to 4.91]

5. Secondary Outcome: Change in Continuous Measure of Quality of Life (QWB)
Description: range - 0-1 (higher score represents greater wellbeing)
Time Frame: Baseline, 6 months
Population: Full sample
Measure: Mean (Standard Deviation); unit: Units on a Scale from 0-1
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 112 | 118
Units on a Scale from 0-1 | -0.00407 (0.1086) | -0.00800 (0.1019)

6. Secondary Outcome: Satisfaction With Care (ECHO)
Description: Using any number from 0 to 10, where 0 is the worst care possible and 10 is the best care possible, what number would you use to rate all the care you received for personal or emotional problems in the last 6 months?
Time Frame: 6 months
Population: Full sample. Data missing for 1 Arm 1 subject and 3 Arm 2 subjects
Measure: Mean (Standard Deviation); unit: 0-10 self reported rating
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 111 | 115
0-10 self reported rating | 8.83423 (1.17964) | 7.7043 (2.2671)

7. Secondary Outcome: Medication Adherence, Defined as Taking Medication <80% of Days
Description: 0 - taking medication <80% of days; 1 - taking medications >=80%
Time Frame: 6 months
Population: Sample only for 205 patients prescribed medications.
Measure: Number; unit: participants
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 104 | 101
participants | 62 | 68
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p = 0.65, Mixed Models Analysis; Odds Ratio, log = 0.86, 95% CI 2-sided [0.46 to 1.62]

8. Secondary Outcome: Received at Least 8 Sessions of Exposure Based Therapy
Description: 0 - received <8 sessions of exposure based therapy; 1 - received >=8 sessions of exposure based therapy
Time Frame: 12 months
Population: Full Baseline Sample
Measure: Number; unit: participants
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Number analyzed (Participants) | 133 | 132
participants | 36 | 7
Statistical Analysis 1: Comparison: Arm 1 Telemedicine Outreach for PTSD vs Arm 2 Treatment as Usual; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 7.9, 95% CI 2-sided [3.2 to 19.6]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Death (Not Study Related). Death was the only adverse event monitored.
Arm/Group | Arm 1 Telemedicine Outreach for PTSD | Arm 2 Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/133 | 5/132
Other Adverse Events (participants affected / at risk) | 0/133 | 0/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Telemedicine Outreach for PTSD (N=133) | Arm 2 Treatment as Usual (N=132)
Death (Not Study Related) (General disorders) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
High enrollment refusal rates may limit external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes